CLINICAL TRIAL: NCT04533789
Title: Wii Sport Games Versus Task-oriented Training on Gait in Children With Unilateral Cerebral Palsy
Brief Title: Virtual Reality versusTask-oriented for Gait in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, Lecturer of physical therapy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/001729
Record Dates: First submitted 2020-08-16; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cerebral Palsy
Keywords: wii sport; task oriented training; hemiplegic cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: G 1 (control) received traditional physical therapy program for 60 min. G 2 (study) received traditional physical therapy program for 30 min. and virtual reality for 30 min.
  G 3 (study) received traditional physical therapy program for 30 min. and task oriented training for 30 min.
  all groups treated for four successive months.
Who Masked: Participant, Investigator
Masking Description: Single (Outcomes Assessor) Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group 1 (control group) and Group 2 (virtual reality group), group 3 (task oriented training)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the control group (Experimental): Group 1 the control group received selected physical therapy program which contain strengthening exercises for upper limb and lower limb muscles, stretching exercises for elbow extensors, hand supinator, wrist extensors, knee extensors and ankle dorsiflexors, balancing exercises, coordination exercises and gait training exercises in open environment.
  Interventions: Other: selected physical therapy program
- virtual reality (Experimental): Group 2 the study group received the same physical therapy program 30 min. plus virtual reality for 30 min.
  Interventions: Other: selected physical therapy program
- Task oriented (Experimental): Group 3 the study group received the same physical therapy program 30 min. plus task oriented training for 30 min.
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Other: selected physical therapy program — strengthening muscles of upper and lower limbs, balancing exercise, gait training in open environment, stretching for elbow flexors and forearm pronators,lower limb hip flexors and knee extensor and ankle dorsiflexors

SUMMARY:
The children with hemiplegic cerebral palsy had a longer gait cycle, slower walking speed, and longer support phase than did the healthy children. The support phase was longer than the swing phase in the children with hemiplegic cerebral palsy

DETAILED DESCRIPTION:
This research aims to evaluate the effect of virtual reality (VR) games on balance recovery of children with cerebral palsy (CP) by quantitatively synthesizing the existing literature, and to further determine the impact of VR game intervention (the duration of each intervention, intervention frequency, intervention cycle, and total intervention time) on the balance recovery of children with CP.

A high-intensity task-oriented training programme designed to improve hemiplegic gait and physical fitness was feasible in the present study and the effectiveness exceeds a low intensity physiotherapy-programme in terms of gait speed and walking capacity in hemiplegic cp. In a future study, seems appropriate to additionally use measures to evaluate physical fitness and energy expenditure while walking.

ELIGIBILITY:
Inclusion Criteria:

1. Their age will ranging from 7 to 9 years.
2. Children participated in this study will from both sexes.
3. Their degree of spasticity will ranged from mild to moderate according to Modified Ashworth Scale.
4. All children will able to walk supported or unsupported by the therapist.
5. Children will able to follow the instructions during testing and training.
6. All children had no fixed contractures or deformities at the lower limb.

Exclusion Criteria:

1. Children with visual or auditory problems.
2. Children with history of epilepsy.
3. Children with structural joints deformities of the lower limbs.
4. Children with history of surgical interference in lower limbs less than one year.
5. Children with convulsions and fixed contractures.
6. Uncooperative children.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
cadence (number) | cadence assessed at day 0.
  number of steps in each min.
cadence (number) | cadence assessed at day 90.
  number of steps in each min.
step length of affected side (cm) | step length assessed at day 0.
  distance between the point of initial contact of one foot and the point of initial contact of the opposite foot (cm)
step length of affected side (cm) | step length assessed at day 90.
  distance between the point of initial contact of one foot and the point of initial contact of the opposite foot (cm)
stride length of affected side(cm) | stride length assessed at day 0.
  the distance from the toe of right foot (starting position) to the toe of right foot (ending position), or the heel of right foot (starting position) to the heel of right foot (ending position). (cm)
stride length of affected side(cm) | stride length assessed at day 90.
  the distance from the toe of right foot (starting position) to the toe of right foot (ending position), or the heel of right foot (starting position) to the heel of right foot (ending position). (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Ali, PhD student, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Wang Y. Gait analysis of children with spastic hemiplegic cerebral palsy. Neural Regen Res. 2012 Jul 15;7(20):1578-84. doi: 10.3969/j.issn.1673-5374.2012.20.008. PMID 25657696
- [Background] Patterson KK, Gage WH, Brooks D, Black SE, McIlroy WE. Evaluation of gait symmetry after stroke: a comparison of current methods and recommendations for standardization. Gait Posture. 2010 Feb;31(2):241-6. doi: 10.1016/j.gaitpost.2009.10.014. Epub 2009 Nov 22. PMID 19932621
- [Background] Grasso R, Assaiante C, Prevost P, Berthoz A. Development of anticipatory orienting strategies during locomotor tasks in children. Neurosci Biobehav Rev. 1998 Jul;22(4):533-9. doi: 10.1016/s0149-7634(97)00041-9. PMID 9595566
- [Result] Gatica-Rojas V, Mendez-Rebolledo G, Guzman-Munoz E, Soto-Poblete A, Cartes-Velasquez R, Elgueta-Cancino E, Cofre Lizama LE. Does Nintendo Wii Balance Board improve standing balance? A randomized controlled trial in children with cerebral palsy. Eur J Phys Rehabil Med. 2017 Aug;53(4):535-544. doi: 10.23736/S1973-9087.16.04447-6. Epub 2016 Nov 24. PMID 27882910

DOCUMENTS (1):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04533789/Prot_000.pdf